CLINICAL TRIAL: NCT01353859
Title: An Open Label, Local, Multicenter , Phase IIIb Interventional Study to Assess the Efficacy of Tocilizumab (TCZ) in Combination With Methotrexate (MTX) in Indonesian Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Non-biologic DMARDs
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Non-biologic DMARDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25536
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: methotrexate

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks for a total of 6 infusions
Drug: methotrexate — 10-25 mg orally weekly

SUMMARY:
This multicenter, open-label, single arm study will assess the safety and efficacy of RoActemra/Actemra (tocilizumab) in combination with methotrexate in patients with active rheumatoid arthritis who have an inadequate response to non-biologic disease-modifying antirheumatic drugs (DMARDs). Patients will receive RoActemra/Actemra 8 mg/kg intravenously every 4 weeks for a total of 6 infusions plus methotrexate 10-25 mg orally weekly. Anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe active rheumatoid arthritis (RA) of >/= 6 months duration
* Prior treatment with DMARDs for >/= 12 weeks (at stable dose for >/= 8 weeks)
* Inadequate clinical response to stable dose of non-biologic DMARD (either single or in combination)

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following enrollment
* Autoimmune disease other than RA
* History of or current inflammatory joint disease other than RA
* Previous treatment with any biologic drug that is used in the treatment of RA
* Intra-articular or parenteral corticosteroids within 6 weeks prior to baseline
* Impaired liver, renal or hematologic function
* Active current or history of recurrent infection
* History of or currently active primary or secondary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Indonesia (5):
  - Bandung
  - Central Jakarta
  - East Java
  - Malang
  - Yogyakarta

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab + Methotrexate (MTX): Participants received tocilizumab 8 milligrams per kilogram (mg/kg) (minimum dose 480 mg, maximum dose 800 mg), intravenously (IV), once every 4 weeks (maximum number of infusions received was 6) and MTX, 10-25 mg per week, at a stable dose; the dose and route of administration of MTX at entry in the study was to be continued without change while on study unless an adjustment was necessary for safety reasons. All participants treated with MTX received either folic acid or leucovorin according to the manufacturer's recommendations.
Period: Overall Study
Arm/Group | Tocilizumab + Methotrexate (MTX)
Started | 39
Completed | 35
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population: all participants included in the study who received at least one dose of study medication. Participants prematurely withdrawn from the study will be considered as nonresponders at the end of the study in all analyses of treatment response variables.
Groups:
- Tocilizumab + MTX: Participants received tocilizumab 8 mg/kg (minimum dose 480 mg, maximum dose 800 mg), IV, once every 4 weeks (maximum number of infusions received was 6) and MTX, 10-25 mg per week, at a stable dose; the dose and route of administration of MTX at entry in the study was to be continued without change while on study unless an adjustment was necessary for safety reasons. All participants treated with MTX received either folic acid or leucovorin according to the manufacturer's recommendations.
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 53 [19 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Low Disease Activity Score
Description: Disease Activity Score using 28-Joint Count (DAS28) was calculated from the number of swollen joints and tender joints using the 28-joint count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and global health assessment (participant-rated global assessment of disease activity using 10-mm visual analog scale [VAS]); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 less than or equal to (≤3.2) equals (=) low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Week 24
Population: ITT population: All participants randomized in the study who received administration of at least one dose of the study drug and who had the last week 24 assessment performed.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 35
percentage of participants | 100

2. Secondary Outcome: Time to Achieve Low Disease Activity (DAS28 ≤3.2)
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 ≤3.2 = low disease activity; time to low disease activity was calculated as the time in weeks from the date of first infusion to the first achievement of DAS28 ≤3.2
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
weeks | 9.5 (5.3)

3. Secondary Outcome: Percentage of Participants With a Clinically Significant Improvement in DAS28 Score
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity; a clinically significant improvement in DAS28 score was defined as a reduction of at least 1.2 units.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
percentage of participants
  Week 4 | 87.2
  Week 8 | 91.9
  Week 12 | 94.7
  Week 16 | 97.3
  Week 20 | 97.3
  Week 24 | 100

4. Secondary Outcome: Time to Clinically Significant Improvement in DAS28
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity; a clinically significant improvement is a reduction in DAS28 score of at least 1.2 units. Time to clinically significant improvement was determined in weeks from the date of first infusion to the date of first achievement of reduction of 1.2 units in DAS28.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
weeks | 12.5 (6.3)

5. Secondary Outcome: Percentage of Participants Achieving DAS28 Remission (DAS28 <2.6)
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. Remission was defined as DAS28 <2.6.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
percentage of participants
  Baseline | 0.0
  Week 4 | 20.5
  Week 8 | 36.8
  Week 12 | 44.7
  Week 16 | 59.0
  Week 20 | 74.4
  Week 24 | 82.1

6. Secondary Outcome: Time to Achieve DAS28 Remission (DAS28 <2.6)
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 remission was defined as DAS28 <2.6. Time to achieve remission was calculated in weeks as the time from the date of first infusion to the date of first achieving remission.
Time Frame: Weeks 4, 8, 12, 16, 20 and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
weeks | 4.4 (1.6)

7. Secondary Outcome: Percentage of Participants With DAS28 <3.2 by Visit
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hour) and global health assessment (participant-rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 ≤3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
percentage of participants
  Baseline | 0.0
  Week 4 | 30.8
  Week 8 | 48.7
  Week 12 | 69.2
  Week 16 | 82.1
  Week 20 | 89.7
  Week 24 | 100

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20%, 50%, and 70% Improvement (ACR20, ACR50, or ACR70) Response
Description: ACR20/50/70 response was defined as ≥20%, ≥50%, or ≥70% improvement, respectively, in swollen/tender joint count (66 joints assessed for swelling and 68 joints assessed for tenderness) as well as improvement in at least 3 of the 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the health assessment questionnaire [HAQ]); and acute phase response: C-reactive protein (CRP) or ESR.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
percentage of participants
  ACR20 | 20
  ACR50 | 34
  ACR70 | 34

9. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: Erythrocyte Sedimentation rate was measured in mm/hour and was used to determine the acute phase response. Lower ESR values indicate reduction in disease activity; normal reference range: 0-20 mm/hr.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
mm/hr
  Baseline | 48.1 (26.1)
  Week 4 | 10.7 (13.5)
  Week 8 | 9.1 (10.5)
  Week 12 | 6.3 (4.3)
  Week 16 | 8.3 (8.3)
  Week 20 | 6.6 (4.3)
  Week 24 | 5.8 (3.3)

10. Secondary Outcome: C-Reactive Protein Levels
Description: CRP levels were measured in milligrams/liter (mg/L) and were used to determine the acute phase response. A reduction in CRP levels is considered an improvement; normal reference range ≤10 mg/L.
Time Frame: Baseline, Weeks 4, 8, 12,16, 20, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab + MTX
Number analyzed (Participants) | 39
mg/L
  Baseline | 17.6 (21.6)
  Week 4 | 2.1 (8.5)
  Week 8 | 0.8 (1.9)
  Week 12 | 0.5 (1.0)
  Week 16 | 1.2 (4.4)
  Week 20 | 1.0 (2.6)
  Week 24 | 0.4 (0.3)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the day of baseline evaluation until the end of study at Week 24.
Arm/Group | Tocilizumab + MTX
Serious Adverse Events (participants affected / at risk) | 2/39
Other Adverse Events (participants affected / at risk) | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab + MTX (N=39)
Sepsis (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab + MTX (N=39)
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Odynophagia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 5
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Injection site ecchymosis (General disorders) | 1
Injection site haematoma (General disorders) | 1
Injection site pain (General disorders) | 1
Pain (General disorders) | 1
Hepatic enzyme increased (Investigations) | 12
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Cold (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Influenza (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Fungal infection (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Azotaemia (Renal and urinary disorders) | 1
Headache (Nervous system disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Pelvic inflammatory disease (Reproductive system and breast disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Pain ankle (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Weakness (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.